CLINICAL TRIAL: NCT03798743
Title: Single Center, Single Arm Phase II Study on Efficacy Evaluation and Bio-marker Analysis of Sintilimab Combined With Docetaxel for Double Platinum-based Chemotherapy Failure Advanced Non-small Cell Lung Cancer
Brief Title: Phase II Study on Sintilimab Combined With Docetaxel for Chemotherapy Failure Advanced NSCLC: the SUCCESS Study
Acronym: SUCCESS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hunan Province Tumor Hospital (Other)
Responsible Party: Principal Investigator, Yongchang Zhang, Professor, Hunan Province Tumor Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SUCCESS
Record Dates: First submitted 2019-01-05; First posted 2019-01-10 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-03

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Non-small Cell Lung Cancer; Sintilimab; Docetaxel
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Docetaxel

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sintilimab Combined With Docetaxel (Experimental): Sintilimab Combined With Docetaxel for Double Platinum-based Chemotherapy Failure Advanced Non-small Cell Lung Cancer
  Interventions: Drug: Sintilimab Combined With Docetaxel

INTERVENTIONS:
Drug: Sintilimab Combined With Docetaxel — Sintilimab 200mgi.v q3w Docetaxel 75mg/m2 i.v q3w
  Other Names: SCD

SUMMARY:
The study aim to Evaluate the combination of ididilimumab and docetaxel alone in the treatment of previous platinum-containing double-drug chemotherapy according to RECIST 1.1Objective remission rate of advanced or metastatic non-small cell lung cancer with negative, driving gene negative (EGFR, ALK, ROS1); (ORR).

DETAILED DESCRIPTION:
This study is a single case of syndilizumab plus docetaxel monotherapy in a Chinese-negative late-stage or metastatic non-small cell lung cancer (NSCLC) failed platinum-containing dual-drug chemotherapy. Center, single arm phase II study. In this study, 30 patients with advanced or metastatic non-small cell lung cancer who had failed platinum-containing dual-drug chemotherapy were treated with rituximab plus docetaxel every 3 weeks until disease progression and intolerance. Toxicity, withdrawal of informed consent, death or other cessation of treatment as prescribed by the program, whichever occurs first. The primary end point was the ORR based on RECIS 1.1, which was evaluated by the Independent Imaging Review Board (IRRC). The longest treatment time for ididibizumab is 24 months. An interim analysis will be conducted during the course of the study. The results and reports will be provided to the Independent Data Audit Committee (IDMC), which determines whether the trial is valid based on the valid cut-off value of the trial and whether the study data can be submitted in advance. Make recommendations to the sponsor. Prior to the interim analysis, the IDMC charter will be finalized and approved by IDMC and the sponsor. The responsibilities and related procedures of IDMC members will be defined in the IDMC charter.

ELIGIBILITY:
Inclusion Criteria:

* Sign written informed consent before any trial-related processes are implemented
* Age ≥ 18 years old and ≤ 75 years old
* Life expectancy exceeds 3 months
* The investigator confirmed at least one measurable lesion according to the RECIST 1.1 standard
* Histological or cytological diagnosis of NSCLC and stage IIIB/IV stage tumors (according to the International Association for the Study of Lung Cancer)Chest tumor staging manual 8th edition judgment) or in multimodal treatment (radiotherapy, surgical resection or radical chemoradiotherapy local treatment)Subjects with relapse or disease progression after treatment for locally advanced disease.
* Subjects must have previously been treated with a platinum-containing dual chemotherapy (carboplatin or cisplatin) regimen for advanced or metastatic tumorsisease progression occurred during or after the period.

  i) receiving maintenance therapy (referring to treatment with no progress after treatment with a platinum-containing dual chemotherapy regimen) and progress Subjects are eligible for inclusion. Ii) treatment of locally advanced disease with platinum-containing adjuvant, neoadjuvant therapy or radical chemoradiotherapy, and completion of treatment Subjects with tumor recurrence or metastasis within 6 months after treatment are eligible.selected.

Iii) administration of platinum-containing adjuvant, neoadjuvant therapy or radical chemoradiotherapy for treatment of locally advanced disease >6 months laterTumor recurrence, and later progressed during or after treatment of a recurrent tumor with a platinum-based regimen Subjects are eligible for inclusion.

* Patients confirmed by histological specimens who are not eligible for EGFR, ALK or ROS1 targeted therapy (with no tumor) EGFR-sensitive mutations and no evidence of ALK, ROS1 gene rearrangement);
* The Eastern Cancer Cooperative Group (ECOG) has a fitness status score of 0 or 1
* Good hematopoietic function, defined as absolute neutrophil count ≥1.5×109/L, platelet count ≥100×109/L, hemoglobin≥90g/L [no blood transfusion or erythropoietin (EPO) within 7 days] Dependency];
* Good liver function, defined as total bilirubin level ≤ normal upper limit (ULN); patients without liver metastases, Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) levels ≤ 1.5 times ULN, alkaline phosphatase ≤ 2.5 times ULN For patients with recorded liver metastases, AST and ALT levels ≤ 5 times ULN;

Exclusion Criteria:

* Small cell lung cancer
* Currently participating in interventional clinical research treatment, or receiving other research medications within 4 weeks prior to the first dose or Used research equipment;
* Previously received the following treatments: anti-PD-1, anti-PD-L1 or anti-PD-L2 drugs or for another stimulus or association a drug that inhibits T cell receptors (eg, CTLA-4, OX-40, CD137);
* Systemic systemic treatment of Chinese patent medicines or immunomodulatory drugs (including thymosin, interferon, interleukin, except for local use of pleural effusion) with anti-lung cancer indications within 2 weeks prior to the first dose, or before the first dose Major surgical treatment within 3 weeks;
* Pulmonary radiation therapy >30 Gy within 6 months prior to first dose
* Completed palliative radiotherapy within 7 days prior to the first dose

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
ORR (Overall response rate) | Approximately 1 years
  Evaluation of objective response rates in patients with advanced or metastatic non-small cell lung cancer who failed to receive platinum-based dual-drug chemotherapy in response to RECIST 1.1 and in combination with docetaxel and docetaxel

SECONDARY OUTCOMES:
PFS (progression free survival time) | Approximately 1 years
  Assessment of the disease-free progression of the subject according to RECIST 1.1
OS (overall survival time) | Approximately 1 years
  Assess the overall survival of the subject according to RECIST 1.1
DOR (duration of response) | Approximately 1 years
  Assessment of subject's duration of remission according to RECIST 1.1
DCR (disease control rate) | Approximately 1 years
  Assessment of subject's disease control rate according to RECIST 1.1
TTR (time to response) | Approximately 1 years
  Assessment of subject's objective response time according to RECIST 1.1

CONTACTS AND LOCATIONS:
Overall Officials: Yongchang Zhang, MD, Principal Investigator — Hunan Cancer Hospital
Locations (1):
- Hunan Provincal Tumor Hospital, Changsha, Hunan, China

REFERENCES:
- [Derived] Zhang Y, Song L, Zeng L, Xiong Y, Liu L, Zhou C, Yang H, Wang Z, Xia Q, Jiang W, Xu Q, Yang N. Sintilimab plus docetaxel as second-line therapy of advanced non-small cell lung cancer without targetable mutations: a phase II efficacy and biomarker study. BMC Cancer. 2022 Sep 5;22(1):952. doi: 10.1186/s12885-022-10045-0. PMID 36064386